CLINICAL TRIAL: NCT07333664
Title: Standard-of-Care Systemic Therapy With or Without Image-Guided 125I Seed Implantation in Patients With Multiple (6-10) Metastatic Lesions: A Randomized Phase 2 Study
Brief Title: Image-Guided 125I Seed Implantation Plus Standard Systemic Therapy for Patients With Multiple Metastatic Lesions
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Li Min (Other)
Responsible Party: Sponsor-Investigator, Li Min, Vice Director, Jinan Military General Hospital
Organization: Jinan Military General Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 960HP20251220
Record Dates: First submitted 2025-12-19; First posted 2026-01-12 (Actual); Last update posted 2026-01-12 (Actual); Status verified 2026-01

CONDITIONS: Metastatic Solid Tumors
Keywords: Multiple Metastases; lodine-125 Seed Brachytherapy; Image-Guided Therapy
MeSH Terms: interventions — Iodine-125

STUDY DESIGN:
Intervention Model Description: This is a randomized, parallel-assignment interventional study with two treatment arms. Participants are assigned in a 1:1 ratio to receive either standard-of-care systemic therapy alone or image-guided iodine-125 (125I) seed implantation plus standard-of-care systemic therapy.
Masking Description: Due to the interventional nature of iodine-125 (125I) seed implantation, participants and treating clinicians are not blinded to treatment allocation. However, radiologists and nuclear medicine physicians who assess imaging outcomes are masked to treatment assignment, and imaging data are reviewed using anonymized datasets to minimize assessment bias.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Standard-of-Care Systemic Therapy (Active Comparator): Participants receive standard-of-care systemic anticancer therapy according to current clinical guidelines and treating physician discretion.
  Interventions: Other: Standard-of-Care Systemic Therapy
- 125I Seed Implantation plus Standard-of-Care Systemic Therapy (Experimental): Participants receive image-guided iodine-125 (125I) seed implantation to multiple metastatic lesions in combination with standard-of-care systemic anticancer therapy.
  Interventions: Other: Standard-of-Care Systemic Therapy; Procedure: Iodine-125 (125I) Seed Implantation

INTERVENTIONS:
Other: Standard-of-Care Systemic Therapy — Systemic anticancer therapy administered according to current clinical guidelines and treating physician discretion, which may include chemotherapy, immunotherapy, targeted therapy, and/or maintenance therapy.
Procedure: Iodine-125 (125I) Seed Implantation — Image-guided implantation of iodine-125 (125I) radioactive seeds to multiple metastatic lesions for local tumor control, performed under CT guidance (with PET/CT fusion planning when clinically indicated) according to institutional standards.
  Arms: 125I Seed Implantation plus Standard-of-Care Systemic Therapy

SUMMARY:
Patients with more than five and up to ten metastatic lesions often have limited tolerance for surgery, radiotherapy, or thermal ablation because of cumulative treatment burden or expected toxicity. In this setting, systemic therapy alone frequently remains the primary treatment option.

This prospective, open-label, randomized phase 2 study evaluates whether image-guided iodine-125 (125I) seed implantation, when added to standard-of-care systemic therapy, can improve disease control compared with standard systemic therapy alone in patients with multiple metastatic lesions. Clinical outcomes including progression-free survival, overall survival, safety, and quality of life will be prospectively assessed.

DETAILED DESCRIPTION:
This is a prospective, open-label, randomized phase 2 interventional study designed to evaluate the efficacy and safety of image-guided iodine-125 (125I) seed implantation in combination with standard-of-care systemic therapy compared with standard systemic therapy alone in patients with multiple metastatic lesions. Patients with more than five and up to ten extracranial metastatic lesions often have limited tolerance for surgery, radiotherapy, or thermal ablation due to cumulative treatment burden or expected toxicity, and in this setting, systemic therapy alone frequently remains the only treatment option. This study therefore explores the potential role of image-guided radioactive seed implantation as an additional local treatment strategy for this patient population.

After eligibility confirmation and baseline assessments, participants will be randomly assigned in a 1:1 ratio to receive either standard-of-care systemic therapy alone or image-guided 125I seed implantation plus standard-of-care systemic therapy. Randomization will be performed using a predefined allocation scheme, and the study is conducted in an open-label manner due to the interventional nature of the procedure.

The primary endpoint of the study is progression-free survival (PFS), defined as the time from randomization to disease progression or death from any cause, whichever occurs first. Secondary endpoints, aligned with prior randomized studies of metastasis-directed therapy, include overall survival, time to initiation of a new systemic therapy, treatment-related adverse events, and patient-reported quality of life. Exploratory objectives include descriptive analyses of patterns of disease progression.

Participants assigned to the experimental arm will undergo image-guided 125I seed implantation targeting multiple metastatic lesions, performed under CT guidance (with PET/CT fusion planning when clinically indicated) according to institutional standards. Systemic anticancer therapy will be administered in both study arms at the discretion of the treating physician in accordance with current clinical guidelines. All participants will undergo scheduled clinical and imaging follow-up, with disease progression assessed using RECIST version 1.1 and/or PERCIST criteria.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years.
* Histologically or cytologically confirmed malignant solid tumor with metastatic disease.
* Presence of more than five and up to ten (6-10) extracranial metastatic lesions, identified on CT or PET/CT imaging and assessable by RECIST version 1.1 (and/or PERCIST when PET imaging is used).
* At least one metastatic lesion considered suitable for image-guided iodine-125 (125I) seed implantation according to institutional assessment.
* Eastern Cooperative Oncology Group (ECOG) performance status of 0-2.
* Adequate organ function to undergo interventional procedures and systemic therapy, as determined by institutional standards.
* Ability to understand and willingness to provide written informed consent.

Exclusion Criteria:

* Diffuse or unstable central nervous system involvement, including leptomeningeal disease or uncontrolled/symptomatic brain metastases requiring immediate local intervention.
* Medical conditions that preclude safe interventional procedures, including uncontrolled infection, severe cardiopulmonary dysfunction, or other serious systemic illness, as judged by the investigator.
* Contraindications to percutaneous implantation, such as uncorrectable coagulation disorders, high bleeding risk, lack of a safe needle path, or unacceptable risk to critical organs.
* Pregnancy or breastfeeding.
* Inability to provide informed consent or comply with study procedures, due to severe psychiatric illness, cognitive impairment, or other limiting conditions.
* Any other condition that, in the investigator's judgment, would make the patient unsuitable for study participation or compromise patient safety or study integrity.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2026-01 (Estimated); Primary Completion 2027-01-01 (Estimated); Study Completion 2028-01-01 (Estimated)

PRIMARY OUTCOMES:
Progression-Free Survival (PFS) | From randomization up to 12 months
  Progression-free survival is defined as the time from randomization to disease progression or death from any cause, whichever occurs first. Disease progression will be assessed using RECIST version 1.1 and/or PERCIST criteria, based on the baseline imaging modality.

SECONDARY OUTCOMES:
Overall Survival (OS) | From randomization up to 24 months
  Overall survival is defined as the time from randomization to death from any cause.
Time to Initiation of a New Systemic Therapy (TTNT) | From randomization up to 12 months
  Time to initiation of a new systemic therapy is defined as the time from randomization to the start of a new line or regimen of systemic anticancer therapy due to disease progression or clinical decision.
Local Control of Treated Lesions | From intervention up to 12 months
  Local control is defined as the absence of in-field progression of metastatic lesions treated with iodine-125 (125I) seed implantation on follow-up imaging.
Safety and Treatment-Related Adverse Events | From intervention through 12 months
  Incidence and severity of adverse events, including procedure-related toxicities, graded according to the Common Terminology Criteria for Adverse Events (CTCAE).
Quality of Life (QoL) | Baseline, and 6 months
  Quality of life is assessed using the European Organisation for Research and Treatment of Cancer Quality of Life Questionnaire-Core 30 (EORTC QLQ-C30). Scores range from 0 to 100. Higher scores on functioning scales and global health status indicate better outcomes, while higher scores on symptom scales indicate worse symptoms.

OTHER OUTCOMES:
Patterns of Disease Progression | From the date of randomization until the date of first documented disease progression, assessed up to 24 months.
  Patterns of disease progression will be descriptively analyzed, including the development of new metastatic lesions versus progression of pre-existing lesions, based on radiographic and/or clinical assessment at the time of disease progression.

CONTACTS AND LOCATIONS:
Locations (1):
- The 960th Hospital of People's Liberation Army (PLA), Jinan, Shandong, China

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual participant data (IPD) will be made available to qualified researchers upon reasonable request after completion of the study and publication of the primary results. Data to be shared may include demographic information, treatment assignment, key efficacy outcomes, adverse events, and imaging-derived parameters. A data-sharing agreement will be required to ensure appropriate use of the dataset.
Supporting Information: Study Protocol, ICF
Time Frame: Individual participant data (IPD) will be available beginning 6 months after publication of the primary study results and will remain available for 5 years following publication, or until the main study database is closed, whichever occurs first.
Access Criteria: Qualified researchers affiliated with academic institutions or recognized research organizations may request access to de-identified individual participant data (IPD), including imaging-derived parameters, dosimetric results, and clinical outcome data.Requests must include a brief research proposal describing the scientific rationale, objectives, and planned analyses. Approval will be granted by the study's principal investigator and institutional ethics committee. Data will be shared through secure institutional data transfer systems after execution of a formal data sharing agreement that ensures patient confidentiality and compliance with applicable privacy regulations.